CLINICAL TRIAL: NCT05269199
Title: Sexual Health Impact of Using Pre-exposure HIV Prophylaxis
Acronym: SatisPreP
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 JACOMET
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2021-10

CONDITIONS: Pre-exposure HIV Prophylaxis (PrEP)
Keywords: PrEP; MSM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiological and psychosociological survey of people on pre-exposure HIV prophylaxis (PrEP).

DETAILED DESCRIPTION:
This study is perform to study the sexual health satisfaction of men who have sex with men (MSM), since the use pre-exposure HIV prophylaxis (PrEP), compared to the time before PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, male having sex with men, not infected with HIV, and using HIV prophylaxis by pre-exposure treatment (PrEP) for at least 1 year, received in consultation for renewal of this prescription.
* Able to give his non-opposition to participate in the research.
* Affiliation to a social security scheme.

Exclusion Criteria:

* Patient under curatorship/guardianship or safeguard of justice
* Refusal to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who have sex with men
Study Population: men who have sex with men (MSM), using Pre-Exposure HIV Prohylaxis (PrEP)
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Sexual health satisfaction | 1 day during the scheduled consultation
  To study the sexual health satisfaction of men who have sex with men (MSM), since the use of HIV prophylaxis by pre-exposure treatment (PrEP), compared to the time before PrEP.

SECONDARY OUTCOMES:
Sentimental satisfaction | 1 day during the scheduled consultation
  To study the sentimental satisfaction since the use of HIV prophylaxis by treatment before exposure (PrEP), compared to the time before PrEP.
Risky behaviours | 1 day during the scheduled consultation
  To study risky behaviours without, then on PrEP since the use of HIV prophylaxis by treatment before exposure (PrEP), compared to the time before PrEP.
Specific care | 1 day during the scheduled consultation
  Describe the use of specific care during PrEP.
Predictors of satisfaction | 1 day during the scheduled consultation
  Define possible predictors of satisfaction with PrEP.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CH Brioude, Brioude
  - CEGIDD Clermont Ferrand, Clermont-Ferrand
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CH Le Puy en Velay, Le Puy-en-Velay
  - CH Montluçon, Montluçon
  - CH Moulins, Moulins
  - CH Vichy, Vichy

IPD SHARING:
Plan to Share IPD: No